CLINICAL TRIAL: NCT02557451
Title: Subretinal Haematoma in AMD: Randomized Controlled Study of 2 Therapeutic Approaches in the Antiangiogenic Era
Brief Title: Surgery, Tissue Plasminogen Activator, Antiangiogenic Agents and Age Related Macular Degeneration Complications
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: BRON PHRC I 2013
Record Dates: First submitted 2015-09-16; First posted 2015-09-23 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Subretinal Haematoma Linked to AMD
MeSH Terms: interventions — Surgical Procedures, Operative

ARMS (2):
- surgery + antiangiogenic (Experimental): surgery (vitrectomy - air - TPA) with injections of an antiangiogenic
  Interventions: Other: Surgery; Procedure: injections of an antiangiogenic
- intravitreal injection of gas/TPA + antiangiogenic (Experimental): intravitreal injection of gas - TPA with injections of an antiangiogenic
  Interventions: Other: Intravitreal injections of gas; Procedure: injections of an antiangiogenic

INTERVENTIONS:
Other: Surgery
  Arms: surgery + antiangiogenic
Other: Intravitreal injections of gas
  Arms: intravitreal injection of gas/TPA + antiangiogenic
Procedure: injections of an antiangiogenic

SUMMARY:
AMD is a disease of the central retina, a zone that enables fine detail activities (reading, detail…). This central zone of the retina can be affected by a haemorrhagic complication when small abnormal vessels suddenly start to bleed inside the retina. Several therapeutic approaches are currently available even though they have never been truly compared. The study will be proposed to patients who need to be treated for haemorrhage of the macula. A certain number of factors will be evaluated to compare the 2 principal approaches currently used in France: surgery followed by injections of an anti-angiogenic OR intravitreal injections of gas followed by injections of anti-angiogenics. This is a multicentre, randomized controlled trial to compare these 2 therapeutic approaches.

These diametrically opposed approaches have very different consequences for patients and in terms of cost for society. The consequences for patients will be immediately measurable so as to determine the best therapeutic approach in terms of functional recovery and the impact of the disease on quality of life, while taking into account the risks inherent to these 2 treatments. The impact on quality of life of these 2 approaches as well as their consequences - an important factor in this disease, which is a cause of sensory handicap - will provide the ophthalmological community with essential information making it possible to validate one or the other of these methods for the management of these haematomas.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting subretinal haematoma linked to AMD

* Occurring at least14 days before the start of therapy
* With the presence of a component overlying the pigmentary epithelium (PE) on the OCT
* And a diameter greater than two pupillary diameters on the retinal photographs

Patients who have provided oral consent

Patients with National Health Insurance cover

Patients available for monthly follow-up

Patient having an effective contraception for the women old enough to procreate during the treatment and during 6 months which follow his stop.

Exclusion Criteria:

* Subretinal haematoma linked to a cause other than AMD (myopia, angioid streaks…)
* History of subretinal haematoma on the same side
* Cloudy humour making it impossible to photograph the fundus of the eye or carry out angiography
* Component of the haematoma exclusively underlying the pigmentry epithelium
* Haemorrhage without lifting of the retina
* Patients presenting an INR greater than 4, thus contra-indicating surgery
* Patients requiring cataract surgery in the first 3 months of the study
* Patients presenting a contra-indication relative to injection of the antiangiogenic (History of AVC bleeding or unknown origin in the last 6 months or MI in the 3 preceding months)
* Pregnant or breast-feeding woman (the patients do not have to breast-feed during at least 6 months after the administration of the last dose of the antiangiogénique)
* Contraindication in the use of ranibizumab: hypersensitivity in the active ingredient or in one of the excipients, eye infection or périoculaire active or suspected, inflammation intraoculaire active severe, treatments anti-VEGF systematic or eye concomitant,
* Contraindication in the use of bevacizumab: hypersensitivity in the active substance or in one of the excipients, the hypersensitivity in the products of the ovarian cells of Chinese hamster (CHO) or in other antibodies human or humanized recombinants, heavy surgical operation dating less than 28 days, not totally healed surgical wound, history of lung bleeding or hémoptysie
* Contraindication in the use of alteplase: hypersensitivity in the active substance, in the gentamicine (a residue of the present manufacturing process in the state of tracks), or in one of the excipients. As all the thrombolytic agents, contraindication in every case associated to a high hemorrhagic risk (current significant hemorrhagic disorder or during the last six months, hemorrhagic known diathesis, concomitant treatment by oral anticoagulants with effective dose, severe or potentially dangerous, obvious or recent bleeding, histories or suspicion of intra-cranial bleeding, suspicion of sub-arachnoid bleeding or history of sub-arachnoid bleeding bound to an aneurysm, histories of severe lesion of the central nervous system (for example néoplasie, aneurysm, surgical operation intracerebral or intrathecal), recent traumatic external cardiac massage (less than 10 days), delivery, recent draining of a vessel not accessible to the compression (for example draining of the subclavian or jugular vein),severe uncontrolled high blood pressure, bacterial endocarditis, pericarditis, acute pancreatitis, gastrointestinal ulcers documented during the last 3 months, esophageal varices, arterial aneurysm, arterial or venous deformations, neoplasia increasing the hemorrhagic risk, severe hepatic disease, including hepatic insufficiency, cirrhosis, portal hypertension (esophageal varicose veins) and evolutionary hepatitis, surgical operation or important traumas during the last 3 months.
* Contraindication in the use of acetazolamide: hypersensitivity in the acetazolamide or in one of excipients, severe hepatic, renal or suprarenal inadequacies, intolerance in sulphonamide, histories of renal colic, allergy in the wheat (other than the coeliac disease).

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity measured on the ETDRS scale | Change from inclusion at 3 months

SECONDARY OUTCOMES:
Visual acuity measured on the ETDRS scale | At 1 month and 6 months
Area of the scotoma presented by the patient according to the Amsler grid | At 1 month, 3 months and 6 months
Quality of life using the VFQ-25 scale | At 3 months and 6 months
Number of injections of an antiangiogenic at the end of the 6 months of treatment | At 6 months
Number of patients with macular bleeding | At 6 months
Area of hypoautofluorescence using the autofluorescence technique | At 3 and 6 months
Complications rate | At 6 months

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - CHU de BESANCON, Besançon
  - CHU de Bordeaux, Bordeaux
  - CH de COLMAR, Colmar
  - CHI de CRETEIL, Créteil
  - CHU de DIJON, Dijon
  - CHU de GRENOBLE, Grenoble
  - HCL - Hôpital de la Croix-Rousse, Lyon
  - CHR de METZ-THIONVILLE, Metz
  - CH de MULHOUSE, Mulhouse
  - CH de NEVERS, Nevers
  - AP-HP Hôpital Lariboisière, Paris
  - Fondation Ophtalmologique A. de Rothschild, Paris
  - CHU de REIMS, Reims
  - Clinique Mathilde, Rouen
  - NHC de STRASBOURG, Strasbourg
  - CHU de TOULOUSE - Hôpital Purpan, Toulouse
  - CHU de NANCY, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Gabrielle PH, Delyfer MN, Glacet-Bernard A, Conart JB, Uzzan J, Kodjikian L, Arndt C, Tadayoni R, Soudry-Faure A, Creuzot Garcher CP. Surgery, Tissue Plasminogen Activator, Antiangiogenic Agents, and Age-Related Macular Degeneration Study: A Randomized Controlled Trial for Submacular Hemorrhage Secondary to Age-Related Macular Degeneration. Ophthalmology. 2023 Sep;130(9):947-957. doi: 10.1016/j.ophtha.2023.04.014. Epub 2023 Apr 22. PMID 37088447